CLINICAL TRIAL: NCT05043207
Title: A Validation of the UAud System for User-operated Audiometry Testing in a Clinical Setting: A Study Protocol for a Blinded Non-inferiority Randomised Controlled Trial.
Brief Title: A Study Protocol for the Validation of UAud in a Clinical Setting.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Southern Denmark (Other)
Collaborators: Innovation Fund Denmark (Individual); William Demant Fonden (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UAUD
Record Dates: First submitted 2021-08-30; First posted 2021-09-14 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Hearing Loss, Sensorineural; Hearing Impairment, Sensorineural
MeSH Terms: conditions — Hearing Loss, Sensorineural

STUDY DESIGN:
Intervention Model Description: randomised control trial
Who Masked: Participant, Care Provider
Masking Description: The HA fitting procedure will be blinded, so neither the participant, the audiologist, nor the follow up test examiner knows which group the participant belongs to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- uAud (Experimental): Patients which hearing aid is fitted based on the audiometry obtained with user-operated automated audiometry.
  Interventions: Diagnostic Test: uAud
- control (Active Comparator): Patients which hearing aid is fitted based on the audiometry obtained with traditional audiometry.
  Interventions: Diagnostic Test: Traditional audiometry

INTERVENTIONS:
Diagnostic Test: uAud — Patients will receive hearing aid treatment based on an audiometry obtained with an user-operated automated audiometry procedure
  Arms: uAud
Diagnostic Test: Traditional audiometry — Patients will receive hearing aid treatment based on an audiometry obtained with an traditional audiometry procedure
  Arms: control

SUMMARY:
The objective of this study is to validate the User-operated Audiometry (UAud) system for user-operated audiometry in a clinical setting, by investigating if hearing rehabilitation based on UAud is non-inferior to hearing rehabilitation based on traditional audiometry, and whether thresholds obtained with the user-operated version of the Audible Contrast Threshold (ACT) test correlates to traditional measures of speech intelligibility.

DETAILED DESCRIPTION:
The project will focus on the initial examination of patients who are referred for hearing aid treatment. This initial examination consists of an audiometry which is currently conducted manually by an audiologist. However, it is possible to conduct an audiometry as a user-operated self-test by using a computer. The project will test if hearing rehabilitation based on the user-operated audiometry is non-inferior to hearing rehabilitation based on the gold standard of manual audiometry. The project will use several types of patient reported measures as well as objective measurements in the clinic. Research of this type is needed to understand if the quality of the hearing aid treatment is equal no matter the type of examination.

Also, the study will investigate whether thresholds obtained with the user-operated version of the Audible Contrast Threshold (ACT) test correlates to traditional measures of speech intelligibility.

ELIGIBILITY:
Inclusion criteria

* Sensorineural hearing loss with hearing thresholds exceeding 20 dB HL at two or more frequencies in the frequency range of 0.5 to 4 kHz.
* Symmetric hearing loss with a maximum pure-tone average (PTA) (mean of 0.5-1-2-4 kHz) difference between the ears of 15 dB HL.
* Danish native speaker.
* No previous experience with HAs.
* Capable of answering questionnaires through an online mailbox.

Exclusion criteria

* Air-conduction audiometry thresholds exceeding 80 dB HL at two or more frequencies.
* Treatment affected by conductive hearing loss (air-bone gap >10 dB on more than one frequency below 1 kHz).
* Conditions with fluctuating hearing loss, e.g., Menière's, on-going treatment with ototoxic drugs.
* Ear, nose, or throat surgery in the past 12 months.
* Evidence that the participant has made minor use of the HAs during the study (e.g., < 2h per day).
* Visual or motor impairment that might affect the use of the UAud system.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
SSQ12 (Speech, Spatial & Qualities of Hearing scale) | 3 months
  A questionnaire reflecting the patient's subjective assessment of hearing in everyday life.

SECONDARY OUTCOMES:
HINT (Hearing In Noise Test) | 3 months
  A performance test of patients speech intelligibility in noise.

OTHER OUTCOMES:
IOI-HA (International Outcome Inventory for Hearing Aids) | 3 months
  A questionnaire regarding the patient's own perception of hearing aid outcome.
APHAB (Abbreviated Profile of Hearing Aid Benefit). | 3 months
  A questionnaire regarding the patient's own perception of hearing and hearing aid outcome.
HINT-U (Hearing In Noise test - under amplification) | 3 months.
  A variation of the HINT framework targeting potential under amplification of hearing aid sound level.
HINT-O (Hearing In Noise Test - Over amplification) | 3 months.
  A variation of the HINT framework targeting potential over amplification of hearing aid sound level.

CONTACTS AND LOCATIONS:
Overall Officials: Jesper Hvass Schmidt, PhD, Principal Investigator — SDU
Locations (1):
- University of Southern Denmark, Odense, Funen, Denmark

IPD SHARING:
Plan to Share IPD: No
Data is governed by the hospital's GPDR (General Data Protection Regulation) agreements.

REFERENCES:
- [Derived] Pedersen C, Pedersen ER, Laugesen S, Sanchez-Lopez R, Nielsen J, Sorensen CB, Schmidt JH. Comparison of hearing-aid effectiveness based on user-operated versus traditional audiometry: a randomised clinical trial. Int J Audiol. 2024 Dec 2:1-8. doi: 10.1080/14992027.2024.2434897. Online ahead of print. PMID 39620470
- [Derived] Pedersen CC, Pedersen ER, Laugesen S, Sanchez-Lopez R, Nielsen J, Sorensen CB, Sidiras C, Pedersen RG, Schmidt JH. Comparison of hearing aid fitting effectiveness with audiograms from either user-operated or traditional audiometry in a clinical setting: a study protocol for a blinded non-inferiority randomised controlled trial. BMJ Open. 2023 Mar 2;13(3):e065777. doi: 10.1136/bmjopen-2022-065777. PMID 36863737